CLINICAL TRIAL: NCT00449267
Title: Clinical Evaluation of Hydrophobic Foldable Intraocular Lenses
Brief Title: Aurolab Hydrophobic Foldable Intraocular Lens Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aurolab (Other)
Responsible Party: Dr. Haripriya Aravind, Aravind Eye Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1PN1010614
Record Dates: First submitted 2007-03-17; First posted 2007-03-20 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Cataract
Keywords: Lenses, Intraocular; Prospective Studies; Visual acuity; Clinical Trial
MeSH Terms: conditions — Cataract | interventions — Lenses, Intraocular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Intraocular Lens

INTERVENTIONS:
Device: Intraocular Lens — Phacoemulsification with in the bag implantation of the IOL
  Other Names: Aurovue, Model HP757SQ

SUMMARY:
The purpose of this study is to evaluate whether hydrophobic intraocular lenses manufactured by aurolab are safe and effective in the surgical treatment of cataract.

DETAILED DESCRIPTION:
Hydrophobic as the name suggests is fear for water. Hydrophobic foldable IOLs are made from acrylic material. Aurolab has developed its own hydrophobic acrylic material. This material has been subjected to several biocompatibility studies and it has proved itself to be biocompatible.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 65 years
* Senile Cataract
* Posterior Subcapsular Cataract (PSCC)

Exclusion Criteria:

* Obviously debilitated patients
* Cardiac and other serious illness
* Diabetic Patients
* Traumatic cataract
* Complicated cataract
* Congenital cataract
* Drug induced cataract
* Shallow anterior chamber
* Poor mydriasis
* Amblyopia
* Pseudo exfoliation (PXF)
* Dense posterior polar cataract (PPC)
* One eyed patients
* Glaucoma
* Uveitis
* Corneal Pathology
* Retinal Pathology
* Intra operative complications like PC rupture, Zonular dialysis

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 10days, 40 days, 150 days post operatively

SECONDARY OUTCOMES:
Refraction | 10days, 40 days, 150 days post operatively
Intraocular pressure | 10days, 40 days, 150 days post operatively
Corneal status | 10days, 40 days, 150 days post operatively
Iritis | 10days, 40 days, 150 days post operatively
IOL decentration | 10days, 40 days, 150 days post operatively
IOL tilt | 10days, 40 days, 150 days post operatively
IOL discoloration | 10days, 40 days, 150 days post operatively
IOL opacity | 10days, 40 days, 150 days post operatively
Cystoid macular oedema | 10days, 40 days, 150 days post operatively
Hypopyon | 10days, 40 days, 150 days post operatively
Endophthalmitis | 10days, 40 days, 150 days post operatively
Pupillary block | 10days, 40 days, 150 days post operatively
Retinal detachment | 10days, 40 days, 150 days post operatively
Status of anterior and posterior capsule | 10days, 40 days, 150 days post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Haripriya Aravind, MBBS, MS, Principal Investigator — Aravind Eye Hospital, Madurai
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India